CLINICAL TRIAL: NCT06745817
Title: Challenges in Achieving Adequate Dietary Status of Women of Reproductive Age (NutriFem)
Brief Title: Challenges in Achieving Adequate Dietary Status of Women
Acronym: NutriFem
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: National Institute of Public Health, Slovenia (Other Government); VIST - Faculty of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: KEP-4-14/2024; L3-50125 (Other Grant/Funding Number: Slovenian Research And Innovation Agency); L3-50125 (Other Grant/Funding Number: Ministry of Health, Republic of Slovenia)
Record Dates: First submitted 2024-12-04; First posted 2024-12-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Nutritional Status; Nutrient Deficiency; Micronutrient Deficiency; Vitamin D Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Iron-deficiency; Diet; Dermis Density; Dermis Thickness; Skin Elasticity; Body Composition; Physical Activity
Keywords: dietary intake; nutritional status; micronutrients
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Anemia, Iron-Deficiency; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be destroyed after analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1 sample: Adult women (20-49 years) with different dietary habits
  Interventions: Diagnostic Test: Screening questionnaire
- Part 2 sample: Adult women (20-49 years) with different dietary habits invited from Part 1, including also subsamples of vegans, vegetarians, omnivores
  Interventions: Diagnostic Test: Assessement of nutritional status; Diagnostic Test: Dermis density and thickness; Diagnostic Test: Skin elasticity; Diagnostic Test: Body composition measurement; Diagnostic Test: Screening questionnaire

INTERVENTIONS:
Diagnostic Test: Assessement of nutritional status — Assessment of socio-demographic parameters, anthropometric and body composition parameters, food intake (dietary recalls, food propensity questionnaire) and nutritional status (blood biomarkers)
  Groups: Part 2 sample
Diagnostic Test: Dermis density and thickness — Dermis density and thickness will be measured using ultrasonography with Cortex DermaLab 20 MHz US probe.
  Groups: Part 2 sample
Diagnostic Test: Skin elasticity — Skin elasticity will be measured using Cortex DermaLab elasticity probe.
  Groups: Part 2 sample
Diagnostic Test: Body composition measurement — Body composition will be measured using Biostat Multiscan 5000.
  Groups: Part 2 sample
Diagnostic Test: Screening questionnaire — Screening questionnaire: assessment of socio-demographic parameters, use of food supplements, health status, dietary habits

SUMMARY:
The aim of the study is to investigate the dietary habits of women of reproductive age (20-49 years). We aim to obtain epidemiological data on the intake and adequacy of key macronutrients and micronutrients, as well as to explore associations with various health indicators. Additionally, we will focus on the nutritional status of subgroups with specific dietary practices, such as vegetarians and vegans.

DETAILED DESCRIPTION:
Key scientific challenges addressed in this study are to investigate the dietary habits and nutritional status of women of reproductive age, to provide epidemiological data on the nutrient intakes in this group (including intakes of key micronutrients) and investigate their relationship with various markers of health. We will evaluate dietary behaviours and special dietary practices among women of reproductive age in Slovenia, through age-representative sampling approach. We will also detailly assess dietary supplementation practices in this population group. Dietary intakes of macro and key micronutrients and nutritional/health status will be evaluated using a cross-sectional epidemiological study.

Further we will investigate links between dietary behaviours with nutritional and health status in order to identify increased nutritional and health risk, as well as potential benefits of different dietary practices. We will particularly focus into following sub-groups of women: omnivorous women, that do not follow any special diet, women that follow vegetarian diet, and women that follow vegan diet. In order to investigate the status of the key micronutrients, standard blood biomarkers will be used. This will allow us to determine nutritional status for iron, folate, vitamin B12 and vitamin D. Body composition will be estimated using bioelectrical impedance spectroscopy (BIS). Other measurements of health-related parameters will include tissue protein density using ultrasonography.

Study results will give insights into the nutritional status in general group of women of reproductive age and enable us to identify links between dietary behaviours with nutritional as well as health status. Through that approach we will be able to identify potential risk for deficiencies of nutrients in studied population group.

Applying a highly multidisciplinary approach and building on previous research we will address the following:

* evaluate dietary behaviours of women of reproductive age (20-49 years) through representative sampling approach. This will enable identification of diet related risks in this group.
* determine dietary supplementation practices of women of reproductive age (20-49 years). This will allow us to better estimate intakes of specific nutrients, as supplements can be important dietary source of nutrients.
* investigate nutritional status of women of reproductive age (20-49 years) in Slovenia with a combination of validated standard dietary assessment methods and blood biomarkers. This will enable also insights in nutritional status for key micronutrients, including iron, folate, vitamin B12 and vitamin D.
* investigate links between dietary behaviours with nutritional/health status, providing information about sub-populations with higher health risks. To enable this, population of omnivorous subjects will be compared with those on vegetarian and vegan diet.

ELIGIBILITY:
Inclusion criteria:

* Age: 20 to 49 years
* Gender: female
* Agrees to participate in the study (has signed a consent form)

Exclusion criteria:

* Menopause (absence of menstruation for at least 12 months, unless the absence is due to hormonal contraception) or post-menopause
* Pregnancy

Reasons for excluding a participant during the study:

* Inability to participate in the study
* Wishes to discontinue participation
* Incomplete data provided

Additional inclusion criteria for including subpopulations in the second part of the study:

Vegetarians:

* Have followed a vegetarian diet for at least 2 years and do not consume meat or fish more than once a month
* Consume eggs and dairy products more than once a month

Vegans:

- Have followed a vegan diet for at least 2 years and do not consume any animal products more than once a month

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: At least 3,000 women (20-49) from the Central Slovenia will be randomly invited to participate (selection by the Statistical Office of the Republic of Slovenia). We aim for 1,650 responding participants.
  In Part 2, we will include 294 participants from Part 1:
  * 202 women representative of the study population
  * 46 vegetarians and 46 vegans
  To ensure enough participants for Part 2, 550 individuals will be invited. They will be selected using stratified random sampling by age. If needed, we will use the snowball method to recruit more vegetarians and vegans.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of nutrient intake | 1 year
  epidemiology of nutrients intake will be investigated from food records (dietary recalls, food propensity questionaires) [g/day]
Assessment of nutritional deficiencies | 1 year
  epidemiology of nutritional deficiencies will be investigated using blood biomarkers

SECONDARY OUTCOMES:
Assessment of inadequate vitamin D status | 1 year
  epidemiology of vitamin D status will be investigated using serum 25-OH-vitamin D concentration
Assessment of inadequate vitamin B12 status | 1 year
  epidemiology of vitamin B12 status will be investigated using serum vitamin B12 concentration
Assessment of inadequate folate status | 1 year
  epidemiology of vitamin folate status will be investigated using serum folate concentration
Assessment of inadequate iron status | 1 year
  epidemiology of vitamin folate status will be investigated using serum ferritin concentration
Assessment of body composition | 1 year
  epidemiology of body composition will be investigated using Bioimpedance Spectroscopy (BIS) which measures at 50 frequencies ranging from 5 kHz to 1000 kHz giving values for impedance, resistance and reactance of the tissues (all in Ohms) from which body composition (proportion of lean and fat mass) values are calculated.
Assessment of dermal thickness | 1 year
  epidemiology of dermal thickness will be measured using 20 MHz ultrasonography in micrometers
Assessment of dermal density | 1 year
  epidemiology of dermal density will be measured using 20 MHz ultrasonography as an intensity score 0-100
Assessment of skin elasticity | 1 year
  epidemiology of skin elasticity will be measured using Cortex DermaLab elasticity measurement

OTHER OUTCOMES:
Body mass index (BMI) epidemiology of dietary intake of nutrients and fibre will be investigated from food records [g/day] | 1 year
  Weight and height will be combined to report BMI in kg/m^2 and providing insights into prevalence of overweight/obesity
Physical activity | 1 year
  epidemiology of physical activity levels will be investigated using International Physical Activity Questionnaire (IPAQ) - Short Form
Muscle strength | 1 year
  Muscle strength will be measured as grip strength using dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Katja Zmitek, PhD, Study Chair — Nutrition Institute, Ljubljana
Locations (3):
- Slovenia (3):
  - National Institute of Public Health, Slovenia, Ljubljana
  - Nutrition Institute, Ljubljana, Ljubljana
  - VIST Fakulteta za aplikativne vede Zmitek, Ljubljana

IPD SHARING:
Plan to Share IPD: No